CLINICAL TRIAL: NCT03861013
Title: Reward Under Stress: Psychobiological Mechanisms of Resilience to Stress
Brief Title: Reward Under Stress: Effects of a Multidimensional Stress Prevention Program in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chantal Martin Soelch (Other)
Collaborators: University of Fribourg (Other); University of Bern (Other)
Responsible Party: Sponsor-Investigator, Chantal Martin Soelch, Professor, University of Fribourg
Organization: University of Fribourg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Reward_Stress; Project 6239 (Other: FUTURA. University of Fribourg)
Record Dates: First submitted 2018-12-23; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Stress, Psychological
Keywords: Stress management; Intervention program; University students; Perceived stress; Mental health; Anxiety; Depression; Quality of life; Sense of coherence; Self-efficacy; Social support; Resilience; Psychological resources; Reward; Cortisol; Ambulatory assessment
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants were randomized assigned to the intervention group or the wait-list control group. The measurements were taken at the same time for both groups: before and after the intervention, and two follow-up ( at 3 and 6 months)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participation in a multidimensional stress prevention program (GeDStress).
  Interventions: Behavioral: Multidimensional stress prevention program (GeDStress)
- Wait-list control group (No Intervention): Participants on the wait-list control group will not receive any treatment between the baseline and last follow-up. After the study has ended, they have the option to participate in the program.

INTERVENTIONS:
Behavioral: Multidimensional stress prevention program (GeDStress) — The multidimensional stress prevention program (GeDStress) is composed of 8 session of 2-hour weekly sessions and integrated cognitive and behavioral strategies, mindfulness-based activities, emotional regulation and social skills exercises. Brief homework activities were given between sessions. The groups were composed by a maximum of 8 students and were led by two trained clinical psychologists.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to investigate the effects of a multidimensional stress prevention program on psychological and physiological indicators among university students.

DETAILED DESCRIPTION:
University students report increased levels of stress in comparison to the general population of the same age, and that may be associated with an increased risk for psychological problems. Depression, anxiety, substance abuse, sleep- and eating problems are often reported by university students. The effectiveness of cognitive, behavioral, and mindfulness interventions focusing on stress prevention among university students was evidenced. However, these programs are generally based on one way to cope with stress. This study is part of a large three-part study and aimed to investigate the impact of a multidimensional stress prevention program on stress, quality of life, psychological and physical indicators, and also psychological resources in university students. The investigators also aimed to study the impact of the intervention on stress and reward experiences in daily life and reward responses under stress in an experimental task.

A randomized controlled trial study was applied to compare pre- and post-outcomes in an experimental group compared to a wait-list control group. Sixty-four university students were randomly distributed in both groups. The experimental group followed an eight-week stress prevention program (GeDStress), integrating cognitive-behavioral strategies with mindfulness-based exercises, emotional regulation strategies, social skills training and assertiveness activities. This program aims at stress reduction and resilience strategies' increase.

The study protocol was accepted by the Ethics Committee of the Cantons of Vaud and Fribourg (Protocol 261/14) and followed the ethical principles of the Declaration of Helsinki (World Medical Association, 2013) and the local regulatory law. Confidentiality was guaranteed and participants could withdraw from the study at any time. All data collected were deidentified with a code. All participants signed the written informed consent.

Before (T1) and after (T2) the participation in the program, both groups participated to a structured interview, which took between 30 and 60 minutes. After that, participants answered well-validated self-reported online questionnaires about their psychological and physical well-being in French. A link with the questionnaires were sent by email and participants had to complete them during the following days. Participants separately received their code number and needed approximately one hour to answer the questionnaires.

At T1 and T2, the students realized also an ambulatory assessment to evaluate their stress and reward experiences in daily life. Participants' stress and reward experience in the daily living environment were assessed five times a day during one week using an adaptation of the Experience Sampling Method (ESM), using an electronic assessment tool. Subjects were asked to report the most important event that happened between the current and the previous measurement and they were then asked to appraise the current situation, their mood, the minor daily events, the related positive and negative affects as well as stress-related experience. In parallel, saliva samples were collected six times a day in order to determine cortisol levels in saliva, to measure the objective level of stress and to combine reported subjective stress with the physiological measures of stress. Saliva samples were obtained by spitting in a tube, and collected saliva samples were stored at -20°C in a deep freeze at the Department of Psychology of the University Fribourg until to be sent to the laboratory for the analysis.

Before and after, the participants also took part in an experimental task to evaluate the reward under stress. The subjects performed the Fribourg reward task developed by Martin-Soelch et al. (2009) to measure reward under a moderate psychological stress. The task comprises two levels of difficulty, which are differentiated through the number of items (3 or 7) to be remembered. The subjects saw first see a fixation cross, followed by the display of the cue about the level of difficulty and whether they can earn money or not during the trial for 1500 ms. After the cue, the subjects saw a fixation cross for 500 ms and then, an array of yellow circles (3 or 7) was displayed for 1500 ms. After a delay, during which a fixation cross was displayed on the screen for 3000 ms, a green circle was presented at any position on the screen for 1500 ms. The subjects had to decide as quickly as possible whether this circle was at the same position as one of the circle presented previously. After the response time has elapsed, the circle disappeared. Half the time, a fixation cross was displayed on the screen for 2000 ms. In the rewarded condition, a feedback about the win and about the cumulated amount of earned money appeared for 1000 ms followed by the balance account for 1000 ms. In the non-rewarded condition, a blank screen was displayed. During the rewarded condition, the subjects could earn a monetary reward. The amount of the monetary reward that could be won varied between two conditions, a low monetary reward consisting in CHF 0.10 or a high monetary reward consisting in CHF 1. The subjects were instructed that they would receive the sum shown at the end of the experiment. The subjects were asked to rate their mood with a visual analog scale in regular intervals. The induction of moderate stress and to evaluate the effects of stress on physiology and brain activation would involve unpredictable mild electric shock induction during the task. At the beginning of each block, the subjects were informed if electric stimulation would be given during the block. In the second block, the electric stimulation can happen at any moment of the trial in an unpredictable fashion for the participant. The intensity of the electric shock was determined before the experiment with each subject individually, to make sure that the intensity of the shock was under the individual pain threshold. In order to measure the level of stress, saliva samples were collected before and after each block (condition), and 10 and 20 minutes after the end of the task, in order to determine cortisol levels in saliva during the different conditions of the task.

Two follow-up sessions were composed by the online self-reported questionnaires, and were measured in both groups at 3 (T3) and 6 (T4) months after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* being older than 18 years old,
* having a good understanding of French or German
* being a student at the University Fribourg

For the other parts of the study:

- being right-handed

Exclusion Criteria:

* the presence of an endocrinological condition,
* history or presence of a neurological disorder or brain injury,
* use of psychotropic drugs,
* presence of a mental disorder, and
* participating in another psychological intervention and participating in the longitudinal part of this study.

For the other parts of the study

- general MRI exclusion criteria, i.e. presence of claustrophobia, being pregnant (tested with a pregnancy test), metal in the body (pacemakers, aneurysm's clips, metallic prosthesis, cochlear implant…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03-14 (Actual); Primary Completion 2017-06-04 (Actual); Study Completion 2017-06-04 (Actual)

PRIMARY OUTCOMES:
Change in depression scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on the Beck Depression Inventory (BDI-II). The BDI-II is a 21-item self-report screening assessing current symptoms of depression. Total score are ranging from 0 to 63. Higher scores indicate severe depressive symptoms.
Change in anxiety trait and state scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on State-Trait Anxiety Inventory (STAI). The STAI is a 40-item inventory designed to assess anxiety levels. Two subscores can be calculated: state and trait anxiety, scores are ranging from 20-80 for each subscore. Higher scores indicate greater anxiety.
Change in sense of coherence scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Sense of Coherence Scale (SOC-13). Sense of coherence is defined as: a global orientation that expresses the extent to which one has a pervasive, enduring though dynamic feeling of confidence that (1) the stimuli deriving from one's internal and external environments in the course of living are structured, predictable, and explicable (comprehensibility); (2) the resources are available to one to meet the demands posed by these stimuli (manageability) ; and (3) these demands are challenges, worthy of investment and engagement (meaningfulness) (Antonovsky, 1987, p.19). This13-item scale measures the sense of coherence, composed of three domains: comprehensibility (scores ranged between 5 and 35), manageability (scores ranged between 4 and 28) and meaningfulness (scores ranged between 4 and 28). A score for each domain and a total score can be obtained by adding the scores. A high total score (ranged between 13 and 91) expresses a stronger sense of coherence.
Change in burnout scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Maslach Burnout Inventory (MBI), student version. This a 27-item inventory that evaluates the frequency of burnout in students. Three subscales can be computed by adding the items: the Emotional Exhaustion (EE) (scores ranging from 0 to 54), the Depersonalization (DP) (scores between 0 and 42), and the Personal Accomplishment (PA) (scores between 0 and 66). Higher scores in EE and DP and low scores in PA expresses higher level of burnout. A total score can also be computed by averaging all items (scores: ranged between 0 and 81). A high total score expresses high level of burnout.
Change in social anxiety scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Liebowitz Social Anxiety Scale (LSAS-SR). It is a 24-item measure assessing social anxiety symptoms severity. Two subscales can be calculated: fear and avoidance of different social situations. A total score can also be calculated by adding the scores obtained in each subscale. Total scores are ranging from 0-144. Higher scores indicated higher levels of social anxiety.
Change in quality of life scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on the World Organization Quality of Life (WHOQOL-BREF). This 26-item version of the WHOQOL assess shortly the quality of life. A global score and four domains: physical (PHYS), psychological (PSYCH), social (SOC) and environmental (ENVIR) quality of life can be computed. The four domains are computed by averaging the items, this score can be multiplied by four to compare with the domains of the WHOQOL-100. The scores are ranged between 0 and 100. Higher scores mean higher perception of quality of life.
Change in difficulties in emotion regulation scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Difficulties in Emotion Regulation Scale (DERS). This brief self-report 36 item questionnaire evaluates multiple aspects of emotion dysregulation. Six subscales can be computed: non acceptance of emotional responses (scores ranging from 1 to 30), difficulties engaging in goal directed behavior (scores ranging from 1 to 25), impulse control difficulties (scores ranging from 1 to 30), lack of emotional awareness (scores ranging from 1 to 30), limited access to emotion regulation strategies (scores ranging from 1 to 40), lack of emotional clarity (scores ranging from 1 to 25). A score total can be obtained by adding the scores of the 6 subscales (scores ranging from 6 to 180), with higher scores indicating higher difficulties in emotion regulation.
Change in perceived stress scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Perceived Stress Scale (PSS). This 14-item scale measures degree to which situations in one's life are appraised as stressful. Higher scores indicate a higher level of perceived stress (scores ranging from 0 to 56).
Change in general self-efficacy scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on the General Self-Efficacy Scale (GSE). This 10-items scale assess the general self-efficacy. A higher score (ranging from 10 to 40) indicates a better general self-efficacy.
Change in mindfulness skills scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Kentucky Inventory of Mindfulness Skills (KIMS). This 39-item self-report questionnaire measures four dimensions : observing (scores ranging from 12 to 60), describing (scores ranging from 8 to 40), acting with awareness (scores ranging from 10 to 50)and accepting without judgment (scores ranging from 9 to 45).
Change in symptoms of mental health scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Scores on Symptom Checklist (SCL-27-plus), a multidimensional screening instrument for mental problems. Composed of 27 items, 5 scales on current symptoms can be evaluated: depressive (scores ranging from 0 to 10), vegetative (scores ranging from 0 to 10), agoraphobic (scores ranging from 0 to 8), and sociophobic symptoms (scores ranging from 0 to 10) and pain (scores between 0 and 12). Each scale is computed by averaging the corresponding items. A global severity index can also be computed by averaging 25 items (score between 0 and 50). A lifetime assessment for depressive symptoms (sum of the items, scores ranged between 5 = possible lifetime depression and 10= no depression) and a screening question for suicidality (sum of 3 items, scores ranged between 3 = risk of suicide and 6 = little or no risk) are also included.
Change in self-compassion scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Self-compassion Scale Short Form (SCS-SF). This 12-item scale evaluates a global score of self-compassion and 6 subscales: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness and Over-Identification. Higher scores indicating greater self-compassion. Each subscale can be computed by calculating the mean of subscale items (scores between 1 and 2, 5). The global score is obtained by computing the grand mean.
Change in perceived social support scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Multidimensional Scale of Perceived Social Support (MSPSS). A 12-item questionnaire designed to evaluate perceived social support from three sources: Family, Friends and Significant others, by doing the mean of the subscale items. A total score can also be computed by averaging all items. Scores are ranged between 1 and 7. Higher scores indicating higher perceived social support.
Change in reward responsiveness scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Reward Responsiveness and Behavioral Inhibition System Scale (RR/BIS). A 15-items self-reporting questionnaire designed to assess the sensitivity to punishment (BIS) and reward (RR). A score is calculated for each of the two scales (RR: scores ranging from 8 to 32; and BIS scores ranging from 7 to 28) by adding the scores of subscale' items. Higher scores indicated higher sensitivity to reward or punishment.
Change in self-esteem scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on Self-esteem Scale (RSES). This 10-item scale evaluates the global self-esteem of an individual (scores ranging from 10 to 40). High scores indicating high self-esteem.
Change in reactions after traumatic events scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Impact of Events Scale (IES). A 15-item scale designed to measure stress reactions after traumatic impact. A score total (ranging from 0 to 75) and 2 subscales: intrusion (ranging from 0 to 35) and avoidance (ranging from 0 to 40) can be computed. High scores indicating higher levels of intrusion and avoidance.
Childhood trauma | Before the treatment
  Score on the Childhood Trauma Questionnaire (CTQ-SF). A 28-item questionnaire designed to assess retrospective child abuse and neglect. 5 dimensions can be computed (scores ranging from 5 to 25): physical abuse, emotional abuse, physical abuse, sexual abuse and emotional neglect. A total score can be computed by adding all items (scores ranging from 25 to 125). A score higher than 5 indicating experiences of maltreatment or abuse in childhood and youth.
Posttraumatic stress | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on the Posttraumatic Stress Diagnostic Scale (PDS). A 49-item self-report measure providing an assessment of all six PTSD's criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). The nature of the event, and their frequency are evaluated with a checklist including potentially traumatizing events (frequency ranging from "never" to "3 times or more"). A symptom severity score can also be computed (scores ranging from 0 to 51). The cut offs for symptom severity rating are 0 no rating, 1-10 mild, 11-20 moderate, 21-35 moderate to severe and >36 severe.
Change in cannabis abuse scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on the Cannabis Abuse Screening (CAST). A 6-item screening for the cannabis abuse or problematic patterns of cannabis use. Score total ranging from 0 to 24. High scores indicating high risk of having a cannabis use disorder.
Change in coping scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment (only cohorts 2, 3 and 4)
  Score of Coping Ways Checklist (WCC). 27-item questionnaire evaluating 3 coping strategies: problem-focused coping (scores ranging from 10 to 40), emotion-focused coping (scores ranging from 9 to 36), and seeking social support (scores ranging from 8 to 32). Subscales scores are computed by adding correspondent items. Higher scores indicate higher use of the coping strategy.
Change in life orientation scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment (only cohorts 3 and 4)
  Score on the Revised Life Orientation Test (LOT-R). 10-item questionnaire evaluating individual differences in generalized optimism versus pessimism. A total score can be computed, ranging from 0 to 24. Higher total scores reflect higher levels of optimism.
Change in smartphone addiction scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment (only cohorts 3 and 4)
  Score on the Smartphone Addiction Scale Short Version (SAS-SV). 10-item questionnaire developed to identify maladaptive behavior associated with smartphones. The scores are ranged from 10 to 60. Higher scores meaning a higher presence of "smartphone addiction".
Change in internet addiction scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment (only cohorts 3 and 4)
  Score on Internet Addiction Test (IAT). A 20-item scale developed to assess internet addiction or problematic internet use. Scores are obtained by adding all the items (ranging from 20 to 100). The higher the score, the greater the problems Internet use causes.
Changes in clients progress through the course of the therapy scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment. At the end of each session: first session, and 1, 2, 3 , 4, 5, 6, and 7 weeks after the first session.
  Score on the Outcome Questionnaire (OQ.45.2). 45-item self-report questionnaire designed for repeated measurement of client progress through the course of therapy and following termination. 3 subscales: Symptom Distress (SD): score ranging from 0 to 100, Interpersonal Relations (IR): score ranging from 0 to 44, and Social Role performance (SR): scores ranging from 0 to 36. A total score can be computed, score ranging from 0 to 180. The higher the score, the more disturbed the individual.

SECONDARY OUTCOMES:
Change in ambulatory assessment scores | Before the treatment, at the end of the treatment (at 2 months)
  Scores in the 67-item ambulatory assessment. It evaluates stressful situations and their effects on daily life. Items can be evaluated alone or combined in some indicators: context information; mood (scores 1-8; valence, energic arousal, calmness); affective states (positive/negative: mean, scores: 1-7); subjective stress (scores 0-9); daily hassles (positive/negative events, frequency : 1-7); perceived support (mean, scores: 1-7. Be appreciated, understood and perceived support); psychological needs: autonomy, competence, and relatedness (mean, scores: 0-6. General score); activity appraisal (scores: 1-7, 0-9. Stress- or event-related score); activity/events appraisal (scores: 0-7. Dimensions: control, novelty and skill); reward experiences (criticism or compliments. Reward expectation: extrinsic, introjected, identified, and intrinsic); emotion regulation (reappraisal and expressive suppression); thoughts; coping strategies; engagement in pleasant activities; and self-esteem.
Change in the answer to the reward task scores | Before the treatment, at the end of the treatment (at 2 months)
  Scores on the laboratory reward task under stress. The Fribourg reward task is a spatial delayed response task to measure reward under stress, with two levels of difficulty to be remembered: 3 items (low) and 7 (high). First, an array of yellow circles (3 /7) are displayed, then one green circle is presented, and participants have to decide as quickly as possible whether this circle is at the same position as one of the previous circles. Reward is also evaluated by two conditions, participants receive money or not during the trial (non-reinforced or reinforced trials). The amount varies between 2 conditions: low (CHF 0.10) or high reward (CHF 1) (up to CHF 52.80). Participants perform the task twice, in the first (control condition), no stressor was included, in the second, a moderate stress was induced through the administration of six unpredictable mild electric shocks. Early in each block, participants are informed if electric stimulation is given, and the intensity of the electric
Change in cortisol levels in daily life | Before the treatment, at the end of the treatment (at 2 months)
  Cortisol levels during the ambulatory assessment
Change in cortisol levels in laboratory task | Before the treatment, at the end of the treatment (at 2 months)
  Cortisol levels during the laboratory task under stress

OTHER OUTCOMES:
Score in the socio-Economic Position Index (PSES) | Before treatment
  Socio-Economic Position Index (PSES). This socio-economic position index is composed of 4 items, and is computed using the formula: PSES = age - 6 x LE - 4 x PC + 55 (LE = level of education; PC = Professional category). Scores between meaning the relative socio-economic position with regard to the Swiss population: 1-31= lower class, 36-54= lower middle-inferior class ; 55-67 = middle class; 68-80= Upper middle class; > 80 = Upper class).
Information about relatives | Before treatment
  Family Interview for genetic Studies (FIGS). This interview is a guide for systematically collecting diagnostic information about relatives of participants. The FIGS is composed of three parts: General Screening Questions, the Face Sheet, and the symptom checklists. The most general information is gathered by using the General Screening Questions about all known relatives in the pedigree, regardless of how distantly related. The Face Sheet is for each of the informant's first degree relatives, and also for any affected relatives about whom the informant can provide information. The various symptom checklists are used to ferret out the diagnostic details that help make possible a best estimate diagnosis. There are checklists for these disorders: depression, mania, alcohol/drug abuse, psychosis, and paranoid/schizoid/schizotypal personality.
Handedness | Before treatment
  Edinburgh Handedness Inventory (EHI). 4-item instrument evaluating handedness dominance in everyday activities. Total score ranging from 0 (right hand) to 100 (left hand dominance).
Change in nicotine dependance scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Score on the Fagerström Test for Nicotine Dependance (FTND). 6-item test aiming to evaluate the level of nicotine dependence. A total score is computed, ranging from 0 (low dependence) to 10 (very high dependence).
Change in psychotherapy alliance scores | At the end of each session: first session, and at 1, 2, 3 , 4, 5, 6, and 7 weeks after the first session. Only for the intervention group
  California Psychotherapy Alliance Scale (CALPAS). 24-item self-report questionnaire measuring the therapeutic alliance. A total score and 4 scales can be obtained: patient working capacity (PWC), patient commitment (PC), working strategy consensus (WSC), and therapist understanding and involvement, (TUI): therapist responsiveness and engagement from the patient's perspective. Scores can be computed by doing the mean of items corresponding to each subscale or all the items for the total score. Scores are ranging from 1 to 7. Higher the scores, stronger is the therapeutic alliance.
Change in quality of the group relationship scores | At the end of each session: first session, and at 1, 2, 3 , 4, 5, 6, and 7 weeks after the first session. Only for the intervention group
  Score on the Group Questionnaire (OQ-GQ). 30-item questionnaire that provides information about the quality of the group relationship (perception about the relationship they have with the group-as-a-whole, other members and the leader). 3 subscales: positive bonding, positive working and negative relationship. High scores suggest greater positive bonding, positive working, and negative relationship.
Evaluation of the intervention program | At the last session: 8 weeks after the beginning of the intervention
  Questions evaluating the intervention program. Four questions assess participants' appreciation of the content and application of the strategies seen in the program in everyday life. Scores are ranging from 1 to 5. The higher the score, the more beneficial the program was assessed by participants.
Change in the academic success scores | Before the treatment, at the end of the treatment (at 2 months), at 3 and 6 months after the end of the treatment.
  Questions about academic success, Grades obteined: ranged between 1 and 6. 6 being the maximum grade.
Change in psychopathological disorders | Before the treatment, at the end of the treatment (at 2 months)
  Mini-International neuropsychiatric Interview (M.I.N.I)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Will depend of the guidelines of the journal in which published

REFERENCES:
- [Background] Regehr C, Glancy D, Pitts A. Interventions to reduce stress in university students: a review and meta-analysis. J Affect Disord. 2013 May 15;148(1):1-11. doi: 10.1016/j.jad.2012.11.026. Epub 2012 Dec 13. PMID 23246209
- [Background] Dyrbye LN, Thomas MR, Shanafelt TD. Systematic review of depression, anxiety, and other indicators of psychological distress among U.S. and Canadian medical students. Acad Med. 2006 Apr;81(4):354-73. doi: 10.1097/00001888-200604000-00009. PMID 16565188
- [Background] Deasy C, Coughlan B, Pironom J, Jourdan D, Mcnamara PM. Psychological distress and lifestyle of students: implications for health promotion. Health Promot Int. 2015 Mar;30(1):77-87. doi: 10.1093/heapro/dau086. Epub 2014 Oct 14. PMID 25315646
- [Background] Deasy C, Coughlan B, Pironom J, Jourdan D, Mannix-McNamara P. Psychological distress and coping amongst higher education students: a mixed method enquiry. PLoS One. 2014 Dec 15;9(12):e115193. doi: 10.1371/journal.pone.0115193. eCollection 2014. PMID 25506825
- [Background] Heinen I, Bullinger M, Kocalevent RD. Perceived stress in first year medical students - associations with personal resources and emotional distress. BMC Med Educ. 2017 Jan 6;17(1):4. doi: 10.1186/s12909-016-0841-8. PMID 28056972
- [Background] Martin-Soelch C, Kobel M, Stoecklin M, Michael T, Weber S, Krebs B, Opwis K. Reduced response to reward in smokers and cannabis users. Neuropsychobiology. 2009;60(2):94-103. doi: 10.1159/000239685. Epub 2009 Sep 21. PMID 19776653
- See also: Research projects University of Fribourg — http://admin.unifr.ch/futura/content/projects/6239